CLINICAL TRIAL: NCT04760457
Title: One-piece TiZr Mini Implants With Miniaturized Carbon-based Coating Prosthetic Connection for Mandibular Overdentures: a Factorial, Randomized Clinical Trial Testing the Outcomes of Immediate/Delayed Loading and Flapped/Flapless Surgery
Brief Title: Mandibular Overdentures Retained by Mini Implants: a Clinical Trial Comparing Different Surgical and Loading Protocols
Acronym: SMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Goias (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other); Institut Straumann AG (Industry)
Responsible Party: Principal Investigator, Cláudio Rodrigues Leles, Full Professor, Universidade Federal de Goias
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: PI04011-2019
Record Dates: First submitted 2021-01-27; First posted 2021-02-18 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Edentulous Mouth; Complete Edentulism
Keywords: Overdenture; Mini implant; Flapless surgery; Dental implant; Implant loading protocol
MeSH Terms: conditions — Mouth, Edentulous | interventions — Immediate Dental Implant Loading

STUDY DESIGN:
Intervention Model Description: A factorial experiment of two factors is planned, each with two possible values or "levels", and whose experimental units take on all possible combinations of these levels across all such factors (2×2 factorial design), allowing the study to determine the effect of each factor on the response variable, as well as the effects of interactions between factors on the response variable. The tested factors will be: loading protocol (immediate or delayed), and surgical approach (flapped or flapless), resulting in a factorial experiment with four treatment combinations in total. Hence, the design is denoted a 2² factorial, which identifies the number of factors (n=2) and how many levels each factor has (n=2) there are in the design (2²=4).
Who Masked: Outcomes Assessor
Masking Description: The assessment of longitudinal outcomes will be performed by an assessor blinded to the surgical/loading protocols
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- IL-FLS (Active Comparator): Immediate loading (IL) and Flapless surgery (FLS)
  Interventions: Procedure: Implant placement with flapless surgery; Procedure: Implant immediate loading
- IL-FPS (Active Comparator): Immediate loading (IL) and Flapped surgery (FPS)
  Interventions: Procedure: Implant placement with flapped surgery; Procedure: Implant immediate loading
- DL-FLS (Active Comparator): Delayed loading (DL) and Flapless surgery (FLS)
  Interventions: Procedure: Implant placement with flapless surgery; Procedure: Implant delayed loading
- DL-FPS (Active Comparator): Delayed loading (DL) and Flapped surgery (FPS)
  Interventions: Procedure: Implant placement with flapped surgery; Procedure: Implant delayed loading

INTERVENTIONS:
Procedure: Implant placement with flapped surgery — Four mini implants will be placed reflecting a flap.
  Arms: DL-FPS; IL-FPS
Procedure: Implant placement with flapless surgery — Four mini implants will be placed without reflecting a flap.
  Arms: DL-FLS; IL-FLS
Procedure: Implant immediate loading — Four mini implants will be immediately loaded.
  Arms: IL-FLS; IL-FPS
Procedure: Implant delayed loading — Four mini implants will be loaded after a 6-week healing period.
  Arms: DL-FLS; DL-FPS

SUMMARY:
This study aims to test the combined effects of different loading protocols and surgical approaches on clinical and patient-reported outcome measures (PROMs) following the use of four mini implants for mandibular overdenture retention.

The main study hypotheses are:

1. There are significant improvements in PROMs following implant intervention compared to baseline measures;
2. Immediately loaded mini implants have similar failure rates compared to mini implants receiving a delayed 6-week protocol.
3. Flapless surgery has similar post-insertion outcomes compared to flapped surgery.

DETAILED DESCRIPTION:
This study aims to test the combined effects of different loading protocols and surgical approaches on clinical and patient-reported outcome measures (PROMs) following the use of four mini implants for mandibular overdenture retention.

Main study hypotheses:

1. There are significant improvements in PROMs following implant intervention compared to baseline measures;
2. Immediately loaded mini implants have similar failure rates compared to mini implants receiving a delayed 6-week protocol;
3. Flapless surgery has similar post-insertion outcomes compared to flapped surgery.

Statement of clinical relevance:

Mini implants are an alternative to standard implants for overdentures. They are suitable for insertion in narrow ridges, are less invasive, simpler, less costly, and faster to perform, and are especially advantageous for older and frail patients who would benefit from more conservative and less burdensome treatments. Although previous studies reported favorable outcomes regarding patient oral comfort and function, there is a need for implant/attachment systems with higher predictability on implant survival and retention performance in the long-term. This study aims to provide clinical evidence on the newly developed 2.4mm one-piece TiZr mini implant with a miniaturized carbon-based coating attachment.

Methods:

This is a randomized clinical trial using a factorial design, to test the effectiveness of a mandibular overdenture retained by four mini implants. Participants will be randomized using a 2×2 factorial design: immediate/delayed loading (factor 1) and flapless/flapped surgery (factor 2). New conventional complete dentures will be provided as the baseline treatment. Next, eligible participants will be those who completed a 6-month period of denture usage, and are in need of implants to improve the function of the mandibular denture. Imaging exam should present a minimum of 5.4 mm of ridge width in the interforaminal region (recommended for flapless surgery).

Included subjects to take part in the RCT will be randomized to the treatment groups according to the combined study factors - loading protocols: immediate (IL) or delayed (DL); and surgical approaches: flapless (FLS) or flapped (FPS) surgery. Hence, the combined factors will results in four groups:

* IL/FLS (Group I)
* IL/FPS (Group II)
* DL/FLS (Group III)
* DL/FPS (Group IV) Considering the patient's perspective this study design assumed a "worst" protocol (delayed and flapped - Group IV) and a "best" protocol (flapless and immediate - Group I) and two other intermediary conditions (flapped/immediate and flapless/delayed).

All participants will receive four Straumann® Mini Implant System (one-piece Tissue Level implants) with an Optiloc® prosthetic connection and PEEK matrix inserts. Surgery will follow the workflow for the surgical procedure for the Straumann® Mini Implant System concerning preoperative planning, implant bed preparation and implant insertion. For the prosthetic procedures, we will perform a chairside incorporation of the retentive inserts to convert the existing well-fitting and well-functioning lower denture into an overdenture with the Optiloc® Retentive System/Straumann® Mini Implants.

Outcomes will include short-term outcomes (Patient perceived burdens in surgery, postoperative swelling and pain, consumption of analgesics and surgical time) and long-term - 1-year (implant survival and success, peri-implant marginal bone level changes, PROMs, retention force, prosthodontic events) outcomes. Sample size calculation resulted in a total of 74 participants, 18 in each of the four groups. Data analysis will include descriptive and bivariate analyses, Kaplan-Meier curves and regression models using Generalized Estimating Equations (GEE) for longitudinal data.

ELIGIBILITY:
Inclusion Criteria:

* No contraindications for implant surgery (mainly related to uncontrolled systemic diseases);
* Enough bone height in the interforaminal area for an implant length of at least 10 mm;
* Ability to understand and answer the questionnaires used in the study and agree to participate by providing a written informed consent.

Exclusion Criteria:

* Noncompliant participants;
* Disagreement to be randomly allocated to the treatment study groups;
* Signs of untreated temporomandibular disorders or uncontrolled systemic or oral conditions that require additional treatments.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Patient-perceived burdens | Twenty-four hours after implant surgery.
  The Burdens in Oral Surgery Questionnaire (BiOS-Q) will be used to assess patient-perceived burdens. It includes 16 items concerning all aspects of procedures occurring during a surgery. Responses for each item are assessed using a visual analogue scale (VAS) ranging from 0 = no expression of the attribute (e.g. not unpleasant at all) to 100 = maximum expression (e.g. very unpleasant).
Implant survival and success | Incidence thoughout the 12-month follow-up after implant placement.
  Each implant will be assessed according to the health scale of the International Congress of Oral Implantologists (ICOI-Pisa health scale). After clinical assessment, each implant will be classified as 'success', 'satisfactory survival', 'compromised survival' or 'failure'.
Postoperative pain and discomfort | Assessed 24 hours after implant placement.
  A 100-cm graduated visual analog scale will be used to evaluate participants' assessments of pain and discomfort regarding the surgical process. Each participant will indicate their level of pain and discomfort with each parameter by marking a point along the scale.
Postoperative pain and discomfort | Assessed 72 hours after implant placement.
  A 100-cm graduated visual analog scale will be used to evaluate participants' assessments of pain and discomfort regarding the surgical process. Each participant will indicate their level of pain and discomfort with each parameter by marking a point along the scale.
Postoperative pain and discomfort | Assessed 1 week after implant placement.
  A 100-cm graduated visual analog scale will be used to evaluate participants' assessments of pain and discomfort regarding the surgical process. Each participant will indicate their level of pain and discomfort with each parameter by marking a point along the scale.
Consumption of analgesics | Assessed until 1 week after implant placement.
  The number of analgesics consumed by the participant during the post-operative and healing period will be recorded in the patient's file.
Patient Satisfaction | Assessed at baseline (before implant surgery)
  The McGill Denture Satisfaction Instrument - DSI (Awad & Feine, 1998; de Grandmont et al., 1994) will be used to assess patients' satisfaction relating to their prostheses. This is a treatment-specific patient-based outcome assessing satisfaction relating to several aspects of the mandibular prosthesis, including general satisfaction, comfort, stability, aesthetics, chewing ability (ease of chewing), chewing efficiency (ability to crush food in small particles), ease of cleaning, ability to speak and oral condition (condition of their mouth, which can refer to oral health status and was measured by "In general, are you satisfied with your oral condition?''. The subjects will answer on a 100 mm visual analogue scale (VAS) anchored by the words 'not at all satisfied' and 'extremely satisfied'.
Patient Satisfaction | Assessed at the 3-month follow-up visit after implant placement.
  The McGill Denture Satisfaction Instrument - DSI (Awad & Feine, 1998; de Grandmont et al., 1994) will be used to assess patients' satisfaction relating to their prostheses. This is a treatment-specific patient-based outcome assessing satisfaction relating to several aspects of the mandibular prosthesis, including general satisfaction, comfort, stability, aesthetics, chewing ability (ease of chewing), chewing efficiency (ability to crush food in small particles), ease of cleaning, ability to speak and oral condition (condition of their mouth, which can refer to oral health status and was measured by "In general, are you satisfied with your oral condition?''. The subjects will answer on a 100 mm visual analogue scale (VAS) anchored by the words 'not at all satisfied' and 'extremely satisfied'.
Patient Satisfaction | Assessed at the 6-month follow-up visit after implant placement.
  The McGill Denture Satisfaction Instrument - DSI (Awad & Feine, 1998; de Grandmont et al., 1994) will be used to assess patients' satisfaction relating to their prostheses. This is a treatment-specific patient-based outcome assessing satisfaction relating to several aspects of the mandibular prosthesis, including general satisfaction, comfort, stability, aesthetics, chewing ability (ease of chewing), chewing efficiency (ability to crush food in small particles), ease of cleaning, ability to speak and oral condition (condition of their mouth, which can refer to oral health status and was measured by "In general, are you satisfied with your oral condition?''. The subjects will answer on a 100 mm visual analogue scale (VAS) anchored by the words 'not at all satisfied' and 'extremely satisfied'.
Patient Satisfaction | Assessed at the 12-month follow-up visit after implant placement.
  The McGill Denture Satisfaction Instrument - DSI (Awad & Feine, 1998; de Grandmont et al., 1994) will be used to assess patients' satisfaction relating to their prostheses. This is a treatment-specific patient-based outcome assessing satisfaction relating to several aspects of the mandibular prosthesis, including general satisfaction, comfort, stability, aesthetics, chewing ability (ease of chewing), chewing efficiency (ability to crush food in small particles), ease of cleaning, ability to speak and oral condition (condition of their mouth, which can refer to oral health status and was measured by "In general, are you satisfied with your oral condition?''. The subjects will answer on a 100 mm visual analogue scale (VAS) anchored by the words 'not at all satisfied' and 'extremely satisfied'.
Oral health-related quality of life (OHRQoL) | Assessed at baseline (before implant surgery).
  The cross-culturally adapted Brazilian version of the Oral Health Impact Profile for edentulous subjects (OHIP-EDENT) will be used. It contains 19 items divided in four different subscale domains: (I) masticatory discomfort and disability (four items), (II) psychological discomfort and disability (five items), (III) social disability (five items), and (IV) oral pain and discomfort (five items). The items are answerable by a 3-point Likert scale and responses will be summed to result an overall score. Higher scores represent worse OHRQoL.
Oral health-related quality of life (OHRQoL) | Assessed at the 3-month follow-up visit after implant placement.
  The cross-culturally adapted Brazilian version of the Oral Health Impact Profile for edentulous subjects (OHIP-EDENT) will be used. It contains 19 items divided in four different subscale domains: (I) masticatory discomfort and disability (four items), (II) psychological discomfort and disability (five items), (III) social disability (five items), and (IV) oral pain and discomfort (five items). The items are answerable by a 3-point Likert scale and responses will be summed to result an overall score. Higher scores represent worse OHRQoL.
Oral health-related quality of life (OHRQoL) | Assessed at the 6-month follow-up visit after implant placement.
  The cross-culturally adapted Brazilian version of the Oral Health Impact Profile for edentulous subjects (OHIP-EDENT) will be used. It contains 19 items divided in four different subscale domains: (I) masticatory discomfort and disability (four items), (II) psychological discomfort and disability (five items), (III) social disability (five items), and (IV) oral pain and discomfort (five items). The items are answerable by a 3-point Likert scale and responses will be summed to result an overall score. Higher scores represent worse OHRQoL.
Oral health-related quality of life (OHRQoL) | Assessed at the 12-month follow-up visit after implant placement.
  The cross-culturally adapted Brazilian version of the Oral Health Impact Profile for edentulous subjects (OHIP-EDENT) will be used. It contains 19 items divided in four different subscale domains: (I) masticatory discomfort and disability (four items), (II) psychological discomfort and disability (five items), (III) social disability (five items), and (IV) oral pain and discomfort (five items). The items are answerable by a 3-point Likert scale and responses will be summed to result an overall score. Higher scores represent worse OHRQoL.
Prosthodontic maintenance events | Throughout 12 months after overdenture delivery.
  The incidence of prosthodontic repair/adjustment events will be recorded during the clinical assessments.
Surgical time | Procedure (Assessed during the clinical visit of implant placement and overdenture delivery or denture adaptation.)
  The time interval concerning the clinical visit for implant placement and delivery of the overdenture or denture adaptation will me measured and registered.

SECONDARY OUTCOMES:
Masticatory Performance | Assessed at baseline (before implant surgery).
  To perform the masticatory performance test two gums in a dragée form will be used, one blue and one pink, which need to be stuck together manually by wetting them with water and applying moderate force. The participants will be instructed to chew 2 samples of the gum on theirs preferred chewing side for 20 and 50 chewing cycles, respectively, leaving an interval of 1 minute between each chewing sequence.
Masticatory Performance | Assessed at the 3-month follow-up visit after implant placement.
  To perform the masticatory performance test two gums in a dragée form will be used, one blue and one pink, which need to be stuck together manually by wetting them with water and applying moderate force. The participants will be instructed to chew 2 samples of the gum on theirs preferred chewing side for 20 and 50 chewing cycles, respectively, leaving an interval of 1 minute between each chewing sequence.
Masticatory Performance | Assessed at the 6-month follow-up visit after implant placement.
  To perform the masticatory performance test two gums in a dragée form will be used, one blue and one pink, which need to be stuck together manually by wetting them with water and applying moderate force. The participants will be instructed to chew 2 samples of the gum on theirs preferred chewing side for 20 and 50 chewing cycles, respectively, leaving an interval of 1 minute between each chewing sequence.
Masticatory Performance | Assessed at the 12-month follow-up visit after implant placement.
  To perform the masticatory performance test two gums in a dragée form will be used, one blue and one pink, which need to be stuck together manually by wetting them with water and applying moderate force. The participants will be instructed to chew 2 samples of the gum on theirs preferred chewing side for 20 and 50 chewing cycles, respectively, leaving an interval of 1 minute between each chewing sequence.
Maximum voluntary bite force | Assessed at baseline (before implant surgery).
  Maximum voluntary bite force will be measured with a digital gauge (IDDK - Kratos, Cotia, São Paulo, Brazil) in the region of the first molar with three assessments per side.
Maximum voluntary bite force | Assessed at the 3-month follow-up visit after implant placement.
  Maximum voluntary bite force will be measured with a digital gauge (IDDK - Kratos, Cotia, São Paulo, Brazil) in the region of the first molar with three assessments per side.
Maximum voluntary bite force | Assessed at the 6-month follow-up visit after implant placement.
  Maximum voluntary bite force will be measured with a digital gauge (IDDK - Kratos, Cotia, São Paulo, Brazil) in the region of the first molar with three assessments per side.
Maximum voluntary bite force | Assessed at the 12-month follow-up visit after implant placement.
  Maximum voluntary bite force will be measured with a digital gauge (IDDK - Kratos, Cotia, São Paulo, Brazil) in the region of the first molar with three assessments per side.
Peri-implant bone change | Peri-implant bone loss at the 3-month follow-up compared to initial stage (1-week rediograph).
  Periapical radiographs will be obtained and the peri-implant bone level will be measured and compared longitudinally.
Peri-implant bone change | Peri-implant bone loss at the 6-month follow-up compared to initial stage (1-week rediograph).
  Periapical radiographs will be obtained and the peri-implant bone level will be measured and compared longitudinally.
Peri-implant bone change | Peri-implant bone loss at the 12-month follow-up compared to initial stage (1-week rediograph).
  Periapical radiographs will be obtained and the peri-implant bone level will be measured and compared longitudinally.
Bleeding on probing | Assessed at 6-month post-insertion
  Incidence of inflammation of the peri-implant soft tissues
Bleeding on probing | Assessed at 12-month post-insertion
  Incidence of inflammation of the peri-implant soft tissues
Probing depth | Assessed at 6-month post-insertion
  Level of the peri-implant sulcus (in milimiters)
Probing depth | Assessed at 12-month post-insertion
  Level of the peri-implant sulcus (in milimiters)
Suppuration | Assessed at 6-month post-insertion
  Incidence of suppuration on probing the peri-implant soft tissues
Suppuration | Assessed at 12-month post-insertion
  Incidence of suppuration on probing the peri-implant soft tissues

CONTACTS AND LOCATIONS:
Overall Officials: Claudio R Leles, DDS, PhD, Study Director — Universidade Federal de Goias
Locations (1):
- School of Dentistry, Federal University of Goias, Goiânia, Goiás, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Clinical data will be implemented electronically using a dedicated electronic data capturing (EDC) system (REDCap DMS, https://www.project-redcap.org/), hosted by the server infrastructure of the Federal University of Goias. Data will be entered in REDCap using either the web-based application or the REDCap mobile app for iOS/Android. Baseline and longitudinal health-related data, and patient identifying codes used for the analysis will be entered in a REDCap database.
  The Report Builder will be used to create customized reports that are queried in real time.
Supporting Information: Study Protocol
Time Frame: Data will be available after publication of the results in high-impact journals, and until two years hereafter
Access Criteria: Upon request to the study coordinator

REFERENCES:
- [Background] Awad MA, Feine JS. Measuring patient satisfaction with mandibular prostheses. Community Dent Oral Epidemiol. 1998 Dec;26(6):400-5. doi: 10.1111/j.1600-0528.1998.tb01978.x. PMID 9870539
- [Background] de Grandmont P, Feine JS, Tache R, Boudrias P, Donohue WB, Tanguay R, Lund JP. Within-subject comparisons of implant-supported mandibular prostheses: psychometric evaluation. J Dent Res. 1994 May;73(5):1096-104. doi: 10.1177/00220345940730051201. PMID 8006237
- [Background] Demain S, Goncalves AC, Areia C, Oliveira R, Marcos AJ, Marques A, Parmar R, Hunt K. Living with, managing and minimising treatment burden in long term conditions: a systematic review of qualitative research. PLoS One. 2015 May 29;10(5):e0125457. doi: 10.1371/journal.pone.0125457. eCollection 2015. PMID 26024379
- [Background] Enkling N, Saftig M, Worni A, Mericske-Stern R, Schimmel M. Chewing efficiency, bite force and oral health-related quality of life with narrow diameter implants - a prospective clinical study: results after one year. Clin Oral Implants Res. 2017 Apr;28(4):476-482. doi: 10.1111/clr.12822. Epub 2016 Mar 24. PMID 27009835
- [Background] Enkling N, Haueter M, Worni A, Muller F, Leles CR, Schimmel M. A prospective cohort study on survival and success of one-piece mini-implants with associated changes in oral function: Five-year outcomes. Clin Oral Implants Res. 2019 Jun;30(6):570-577. doi: 10.1111/clr.13444. Epub 2019 May 8. PMID 31021481
- [Background] Kanazawa M, Feine J, Esfandiari S. Clinical guidelines and procedures for provision of mandibular overdentures on 4 mini-dental implants. J Prosthet Dent. 2017 Jan;117(1):22-27. doi: 10.1016/j.prosdent.2016.04.020. Epub 2016 Aug 1. PMID 27492988
- [Background] Klein MO, Schiegnitz E, Al-Nawas B. Systematic review on success of narrow-diameter dental implants. Int J Oral Maxillofac Implants. 2014;29 Suppl:43-54. doi: 10.11607/jomi.2014suppl.g1.3. PMID 24660189
- [Background] Leao A, Sheiham A. Relation between clinical dental status and subjective impacts on daily living. J Dent Res. 1995 Jul;74(7):1408-13. doi: 10.1177/00220345950740071301. PMID 7560392
- [Background] Leao A, Sheiham A. The development of a socio-dental measure of dental impacts on daily living. Community Dent Health. 1996 Mar;13(1):22-6. PMID 8634892
- [Background] Lemos CA, Verri FR, Batista VE, Junior JF, Mello CC, Pellizzer EP. Complete overdentures retained by mini implants: A systematic review. J Dent. 2017 Feb;57:4-13. doi: 10.1016/j.jdent.2016.11.009. Epub 2016 Nov 22. PMID 27888049
- [Background] Marcello-Machado RM, Faot F, Schuster AJ, Nascimento GG, Del Bel Cury AA. Mini-implants and narrow diameter implants as mandibular overdenture retainers: A systematic review and meta-analysis of clinical and radiographic outcomes. J Oral Rehabil. 2018 Feb;45(2):161-183. doi: 10.1111/joor.12585. Epub 2017 Dec 2. PMID 29125652
- [Background] Reissmann DR, Semmusch J, Farhan D, Smeets R, Heiland M, Heydecke G. Development and validation of the Burdens in Oral Surgery Questionnaire (BiOS-Q). J Oral Rehabil. 2013 Oct;40(10):780-7. doi: 10.1111/joor.12092. Epub 2013 Aug 27. PMID 24033878
- [Background] Reissmann DR, Enkling N, Moazzin R, Haueter M, Worni A, Schimmel M. Long-term changes in oral health-related quality of life over a period of 5 years in patients treated with narrow diameter implants: A prospective clinical study. J Dent. 2018 Aug;75:84-90. doi: 10.1016/j.jdent.2018.05.019. Epub 2018 May 28. PMID 29852211
- [Background] Schiegnitz E, Al-Nawas B. Narrow-diameter implants: A systematic review and meta-analysis. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:21-40. doi: 10.1111/clr.13272. PMID 30328192
- [Background] Souza RF, Patrocinio L, Pero AC, Marra J, Compagnoni MA. Reliability and validation of a Brazilian version of the Oral Health Impact Profile for assessing edentulous subjects. J Oral Rehabil. 2007 Nov;34(11):821-6. doi: 10.1111/j.1365-2842.2007.01749.x. PMID 17919248
- [Background] Misch CE, Perel ML, Wang HL, Sammartino G, Galindo-Moreno P, Trisi P, Steigmann M, Rebaudi A, Palti A, Pikos MA, Schwartz-Arad D, Choukroun J, Gutierrez-Perez JL, Marenzi G, Valavanis DK. Implant success, survival, and failure: the International Congress of Oral Implantologists (ICOI) Pisa Consensus Conference. Implant Dent. 2008 Mar;17(1):5-15. doi: 10.1097/ID.0b013e3181676059. PMID 18332753
- [Derived] Ferreira de Sa J, Nascimento LN, de Moraes Sousa JF, Curado TFF, Srinivasan M, McKenna G, Schimmel M, Leles CR. The Effect of Implant Distribution on Functional and Patient-Reported Outcomes of Mandibular Overdentures Retained by Four Mini Implants. J Oral Rehabil. 2025 Sep;52(9):1452-1460. doi: 10.1111/joor.14024. Epub 2025 May 9. PMID 40346748
- [Derived] Curado TFF, Nascimento LN, Silva JR, de Paula MS, Schimmel M, McKenna G, Leles CR. Mandibular overdenture retained by four one-piece titanium-zirconium mini implants: A 2-year RCT on patient-reported outcomes. J Dent. 2024 Oct;149:105267. doi: 10.1016/j.jdent.2024.105267. Epub 2024 Jul 26. PMID 39067647
- [Derived] Leles CR, Curado TFF, Nascimento LN, Silva JR, de Paula MS, McKenna G, Schimmel M. Changes in masticatory performance and bite force after treatment with mandibular overdentures retained by four titanium-zirconium mini implants: One-year randomised clinical trial. J Oral Rehabil. 2024 Aug;51(8):1459-1467. doi: 10.1111/joor.13722. Epub 2024 Apr 29. PMID 38685704